CLINICAL TRIAL: NCT05381623
Title: Microvascular Response to the Harvest of Free Gingival Grafts With or Without the Application of Hemostatic Sutures: a Randomized Controlled Clinical Trial Assessing Palatal Blood Flow by Laser Speckle Contrast Imaging
Brief Title: Harvest of Free Gingival Grafts With or Without the Application of Hemostatic Sutures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22/244-EC_X
Record Dates: First submitted 2022-05-13; First posted 2022-05-19 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-06

CONDITIONS: Thin-gingiva; Mucogingival Deformity on Edentulous Ridge; Gingival Recession
Keywords: Connective tissue graft; Free gingival graft; Mucogingival surgery; Mucogingival conditions; Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Allocation to the test or control group will be revealed to the surgeon only after completing the harvest of the free gingival graft.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified suture-less approach (Experimental): Infiltration of local anesthetic (articaine 4% 1:100.000 epinephrine) around the harvesting site and attendance for the establishment of a competent coagulum.
  Interventions: Procedure: Simplified suture-less approach
- Conventional approach (Active Comparator): Application of hemostatic sponges over the donor site and placement of tooth-suspended compressive sutures over the area.
  Interventions: Procedure: Application of hemostatic sponges and compressive sutures

INTERVENTIONS:
Procedure: Simplified suture-less approach — Immediately after the harvest of a free gingival graft from hard palate, at least a half carpule of local anesthetic (articaine 4% 1:100.000 epinephrine) will be infiltrated within the apical border of the harvesting site and another half mesially and distally to the harvesting site. At the end of the mucogingival procedure, the donor site will be evaluated to inquire regarding the presence of a competent coagulum over the wound area. In such a case, no additional procedure will be performed at the recipient site.
  Arms: Simplified suture-less approach
Procedure: Application of hemostatic sponges and compressive sutures — Immediately after the harvest of a free gingival graft from hard palate, hemostatic collagen sponges will be applied over the harvesting site and a series of tooth suspended external mattress sutures (PGA 5/0) will be applied over the area, in order to provide a compressive effect.
  Arms: Conventional approach

SUMMARY:
Randomized, single-center trial with 2 parallel arms and a 1:1 allocation ratio, with the aim of comparing clinical and microvascular healing and patients related outcomes, which follow the harvest of a free gingival graft, where hemostasis has been achieved with either compressive sutures and homeostatic sponges (control) or with a simplified suture-less approach (test).

DETAILED DESCRIPTION:
This randomized two parallel arms controlled clinical trial aims to establish the early microvascular healing, clinical healing, and patients related outcomes, which follow the harvest of a free gingival graft, where hemostasis has been achieved with either compressive sutures and homeostatic sponges (control) or with a simplified suture-less approach (test). The primary outcome is the microvascular healing of the palate14 days after surgery, assessed by measuring the palatal blood flow with a Laser Speckle Contrast Imaging (LSI), expressed in Laser Speckle Perfusion Units (LSPU). Secondary outcomes include the palatal blood flow at 3, 7 and 30 days after surgery, the clinical healing of the palate, the occurrence of postoperative bleeding and patients related outcome measures assessed 14 postoperative days. A figure of 16 subjects per group was obtained based on an expected difference of 7 LSPU, considering a SD of 6.3 SLPU, 80% power, alpha 0.05, and assuming a foreseen drop-out rate of 15%. Patients will be randomly allocated to two groups: test (simplified suture-less approach) and control (compressive sutures and homeostatic sponges). Cases will be the unit of analysis and T-student (normal distribution) or U Mann Whitney (non normal distribution or non parametric variables) will be performed setting the significance level at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (≥ 18 year old), male or female patient from the University Complutense of Madrid, being able to sign an informed consent form, presenting any mucogingival condition requiring the placement of a free gingival graft or a connective tissue graft obtained through the extra oral de-epithelialization of a free gingival graft.

Exclusion Criteria:

* Patients fitting to all the above inclusion criteria will be excluded from the study if unable to attend to the study-related procedures (including the follow-up visits) or if one or more of the following systemic or local exclusion criteria will be found at any time through the study:

Systemic primary exclusion criteria:

1. Compromised general health status contraindicating the study procedures (≥ASA IV);
2. Drug abuse, alcohol abuse, or smoking > 10 cigarettes a day;
3. Chronic use of corticosteroids, NSAIDs, or immune-modulators (any type, any dose);
4. Use of anti-aggregant or anti-coagulant drugs;
5. Pregnant or nursing women;
6. Hypersensitivity to ibuprofen.

Local primary exclusion criteria:

1. History of previous soft tissue surgeries in the area of the harvest;
2. Preoperative evidence of a palate thickness < 2mm in the area of interest;
3. Intraoperative evidence of active bleeding from the harvesting site at the end of surgery, which impedes the stabilisation of a good coagulum over the harvesting area;

Secondary exclusion criteria:

a. Non compliant patients: poor oral hygiene (FMPS >20%) at 2 consecutive visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Palatal microvascular healing | before surgery, 3 days after surgery, 7 days after surgery, 14 days after surgery, 30 days after surgery
  Changes in the palatal blood flow measured with Laser Speckle Contrast Imaging (LSI), expressed in Laser Speckle Perfusion Units (LSPU)

SECONDARY OUTCOMES:
Postoperative bleeding | 14 days after surgery
  Occurrence of postoperative bleeding during the first two postoperative weeks reported by the patients through a dedicated questionnaire
Patients related outcomes measures (PROMS) | 14 days after surgery
  Patients pain and discomfort with respect to the procedure will be evaluated during the first 2 postoperative weeks with a dedicated questionnaire, utilising VAS scales ranging from 0 (no pain) to 10 (maximum pain).
Patients consumption of analgesic rescue medication | 14 days after surgery
  Patients will be asked to report the amount of rescue medication (ibuprofen 600mg) that have assumed for pain control every day during the first 2 postoperative weeks
Wound healing index at the donor site | 7 days after surgery, 14 days after surgery, 30 days after surgery
  Healing at the donor site will be evaluated at 7, 14 and 30 days after the surgery with the wound healing index (WHI) (Huang et al. 2005), using the following criteria: score 1 = uneventful healing with no gingival edema, erythema, suppuration, patient discomfort, or flap dehiscence; score 2 = uneventful healing with slight gingival edema, erythema, patient discomfort, or flap dehiscence, but no suppuration; and score 3 = poor wound healing with significant gingival edema, erythema, patient discomfort, flap dehiscence, or any suppuration. Scoring will be performed by two independent investigators (DP & AD) over clinical pictures.
Wound healing VAS at the donor site | 7 days after surgery, 14 days after surgery, 30 days after surgery
  Healing will be assessed with a VAS scale, scoring 0 in case of evident tissue necrosis and 10 in case of uneventful healing with no signs of edema or erythema.
  Scoring will be performed by two independent investigators (DP & AD) over clinical pictures.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz Alonso, Study Chair — Faculty of Odontology, University Complutense, Madrid, Spain; David Palombo, Study Director — Faculty of Odontology, University Complutense, Madrid, Spain
Locations (1):
- Department of Periodontology, University Complutense Madrid, Spain, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dellavia C, Ricci G, Pettinari L, Allievi C, Grizzi F, Gagliano N. Human palatal and tuberosity mucosa as donor sites for ridge augmentation. Int J Periodontics Restorative Dent. 2014 Mar-Apr;34(2):179-86. doi: 10.11607/prd.1929. PMID 24600654
- [Result] Huang LH, Neiva RE, Wang HL. Factors affecting the outcomes of coronally advanced flap root coverage procedure. J Periodontol. 2005 Oct;76(10):1729-34. doi: 10.1902/jop.2005.76.10.1729. PMID 16253095
- [Result] Molnar E, Fazekas R, Lohinai Z, Toth Z, Vag J. Assessment of the test-retest reliability of human gingival blood flow measurements by Laser Speckle Contrast Imaging in a healthy cohort. Microcirculation. 2018 Feb;25(2). doi: 10.1111/micc.12420. PMID 28976050
- [Result] Sanz-Martin I, Rojo E, Maldonado E, Stroppa G, Nart J, Sanz M. Structural and histological differences between connective tissue grafts harvested from the lateral palatal mucosa or from the tuberosity area. Clin Oral Investig. 2019 Feb;23(2):957-964. doi: 10.1007/s00784-018-2516-9. Epub 2018 Jun 18. PMID 29915931
- [Result] Tavelli L, Barootchi S, Ravida A, Oh TJ, Wang HL. What Is the Safety Zone for Palatal Soft Tissue Graft Harvesting Based on the Locations of the Greater Palatine Artery and Foramen? A Systematic Review. J Oral Maxillofac Surg. 2019 Feb;77(2):271.e1-271.e9. doi: 10.1016/j.joms.2018.10.002. Epub 2018 Oct 11. PMID 30395825
- [Result] Tavelli L, Barootchi S, Greenwell H, Wang HL. Is a soft tissue graft harvested from the maxillary tuberosity the approach of choice in an isolated site? J Periodontol. 2019 Aug;90(8):821-825. doi: 10.1002/JPER.18-0615. Epub 2019 Feb 12. PMID 30690733
- [Result] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963
- [Result] Zucchelli G, Tavelli L, McGuire MK, Rasperini G, Feinberg SE, Wang HL, Giannobile WV. Autogenous soft tissue grafting for periodontal and peri-implant plastic surgical reconstruction. J Periodontol. 2020 Jan;91(1):9-16. doi: 10.1002/JPER.19-0350. Epub 2019 Oct 6. PMID 31461778